CLINICAL TRIAL: NCT01674530
Title: A,Randomized , Double-blind,Double -Dummy Placebo-controlled,Parallel -Group, Multicenter Study to Evaluate the Clinical Equivalence of Lubiprostone 24 mcg Capsules ( Dr. Reddy's Laboratories Ltd.) With AMITIZA® (Lubiprostone ) 24 mcg Capsules ( Sucampo Pharmaceuticals, Inc. ) in the Treatment of Chronic Idiopathic Constipation
Brief Title: Evaluation of Clinical Equivalence Between Two Lubiprostone Products in the Treatment of Chronic Idiopathic Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRL-USG01-L/2012
Record Dates: First submitted 2012-08-21; First posted 2012-08-29 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Idiopathic Constipation
MeSH Terms: interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lubiprostone (Experimental): Manufactured by Dr Reddy's Laboratories Ltd( 24 mcg administered for 7 days )
  Interventions: Drug: Lubiprostone
- AMITIZA® (Active Comparator): Manufactured by Sucampo Pharmaceuticals(24 mcg administered for 7 days)
  Interventions: Drug: Lubiprostone
- Placebo (Placebo Comparator): Manufactured by Dr Reddy's Laboratories Ltd ( 24 mcg adminstered for 7 days )
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lubiprostone — 24 mcg Capsules to be given in the experimental arm with Placebo Of AMITIZA
  Arms: Lubiprostone
Drug: Lubiprostone — 24 mcg Capsules with placebo of Lubiprostone ( Manufactured by Dr Reddy's Laboratories Ltd)
  Arms: AMITIZA®
Drug: Placebo — 24 mcg capsules of both experimental Lubiprostone and AMITIZA
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the clinical equivalence and safety of the test formulation of Lubiprostone 24 mcg capsules manufactured by Dr Reddy's Laboratories Ltd compared to the marketed formulation AMITIZA® ( Lubiprostone) 24 mcg capsules (Sucampo Pharmaceuticals, Inc.) in patients with confirmed Chronic Idiopathic Constipation

DETAILED DESCRIPTION:
Constipation is a common gastrointestinal problem estimated to effect 2-27 % of the population in United States . It is found more commonly in women and elderly . The prevelance of constipation and growing demand for treatment dictate the need for safe and effective treatment options . Lubiprostone is the first chloride channel activator approved by FDA for long term treatment of chronic idiopathic constipation in adult men and women . To provide a generic medicine to the U.S population Dr Reddy's Laboratories intends to conduct this study to evaluate that the Lubiprostone manufactured by it is equally effective and safe as marketed AMITIZA® ( Lubiprostone) 24 mcg capsules (Sucampo Pharmaceuticals, Inc.)

ELIGIBILITY:
Main Inclusion Criteria:

1. Patients who have signed the written informed consent form prior to entering the study.
2. Male or non-pregnant female aged ≥ 18 years with a clinical diagnosis of CIC defined as, on average, < 3 SBMs per week and confirmed by daily diary during the two week baseline/washout period. An SBM is defined as any bowel movement (BM) that does not occur within 24 hours after rescue medication use.
3. Patients with body mass index between 18 and 35kg/m2 (both inclusive)
4. Have one or more of the following symptoms related to BMs for at least 6 months before the baseline visit and confirmed by daily diary during the 2 weeks baseline/washout period:

   i. very hard (little balls) and/or hard stools for at least 25% of the bowel movements ii. sensation of incomplete evacuation following at least 25% of the bowel movements iii. straining at defecation at least a quarter of the time
5. Women of child-bearing potential should have a negative serum pregnancy test prior to beginning therapy and agree to use effective contraceptive methods (at least one medically approved and highly effective method of birth control defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectables, oral contraceptives combined with at least one barrier method, hormonal IUDs, sexual abstinence or vasectomy of the partner) during the study.
6. For patients aged < 50 years, documentation of the results of either a flexible sigmoidoscopy or colonoscopy performed within the five years prior to dosing, showing no mechanical bowel obstruction or organic disorders of the large or small bowel.
7. For patients aged ≥ 50 years, documentation of the results of either a barium enema with flexible sigmoidoscopy or colonoscopy performed within one year prior to dosing, showing no mechanical bowel obstruction or organic disorders of the large or small bowel.

Main Exclusion Criteria:

1. Females who are pregnant, breast feeding, or planning a pregnancy during the proposed study period.
2. Patients of any age with evidence of weight loss, anemia, or rectal bleeding and without documentation of the results of either a flexible sigmoidoscopy or colonoscopy performed during the 6 months prior to dosing.
3. Patients who have documented mechanical bowel obstruction (e.g., bowel obstruction due to tumor, hernia), megacolon/megarectum, or diagnosis of pseudo-obstruction.
4. Patients with known or suspected organic disorders of the large or small bowel (e.g., inflammatory bowel disease, ulcerative colitis, Crohn's Disease) or constipation secondary to a documented cause (e.g., surgery, bowel resection) or acute hernia or with neurologic diseases or other diseases that cause motility problems for example Parkinson's disease and spinal cord injury, etc.
5. Patients with a history of bowel resection.
6. Patients who are regularly using medications, which are known to cause constipation (anticholinergics, narcotics, calcium channel blockers, tricyclic antidepressants, colchicine, iron supplements, magnesium supplements).
7. Patients who are hospitalized for any gastrointestinal or abdominal surgical procedure during the three months prior to dosing.
8. Patients with clinically significant cardiovascular, liver, lung, neurologic, renal or psychiatric disorder, or clinically significant laboratory abnormalities (if laboratory values exceed 2X Upper Limit of Normal the approval of medical monitor should be taken into consideration before randomizing the patient).
9. Use of systemic antibiotics within four weeks prior to baseline.
10. Any current or planned significant change in diet during the study.
11. Participation in a study with any investigational medication within the past 30 days before screening for this study or previous participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 909 (Actual)
Dates: Start 2012-10; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Primary Analysis | Day 8
  Clinical equivalence of the Test and Reference treatments and the superiority of each active treatment over the Placebo in the change from baseline in mean number of SBM's during the 7 day treatment period of the study

OTHER OUTCOMES:
Safety Analysis | Day 8
  The type , frequency and severity of adverse events across the treatment groups will be analyzed at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Ashis Patnaik, M.D, Study Director — Dr. Reddy's Laboratories Limited; Shilpi Dhawan, M.D, Study Director — Dr. Reddy's Laboratories Limited
Locations (92):
- United States (92):
  - Radiant Research, Birmingham, Alabama
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Clinical Research Associates, Huntsville, Alabama
  - Drug Research Group, LLC, Mobile, Alabama
  - Radiant Research, Scottsdale, Arizona
  - Adobe Clinical Research , LLC, Tucson, Arizona
  - Visions Clinical Research, Tucson, Arizona
  - SC Clinical Research, Inc, Tucson, Arizona
  - Preferred Research Partners, Little Rock, Arkansas
  - Anaheim Clinical Trials, Anaheim, California
  - Diagnamics Inc,477 N. El Camino Real,Suite A100, Encinitas, California
  - Advanced Medical Research Institute, Fresno, California
  - Research Center of Fresno, Fresno, California
  - Translational Research Group, North Hollywood, California
  - Staywell Research, Northridge, California
  - Elias Research Associates, Orange, California
  - Benchmark Research, Sacramento, California
  - Medical Center for CR, San Diego, California
  - Shawn K Hassler, San Francisco, California
  - SC Clinical Research, Inc ,1060 E. Foothill Blvd, Suite 204, Upland, California
  - Progressive Clinical Research, Vista, California
  - Horizons Clinical Research Center, Denver, Colorado
  - Radiant Research, Denver, Colorado
  - Lynn Institute of Denver, Denver, Colorado
  - Consultants of Clinical, Boynton Beach, Florida
  - PAB Clinical Research, Brandon, Florida
  - Elite Trials, Clearwater, Florida
  - Health Care Family Rehabilitation and Research Center, Hialeah, Florida
  - Medical Research Unlimited, LLC, Hialeah, Florida
  - Health Awareness ,Inc, Jupiter, Florida
  - Sunrise Medical Research, Lauderdale Lakes, Florida
  - San Marcus Research Clinic, Miami, Florida
  - Pharmax Research Clinic, Miami, Florida
  - Community Research Foundation , Inc., Miami, Florida
  - Florida International Research, Miami, Florida
  - Columbus Clinical Services, Miami, Florida
  - South Medical Research Group , Inc, Miami, Florida
  - Pharma Research International, Inc, Naples, Florida
  - Compass Research, Orlando, Florida
  - Ormond Medical Arts Pharmaceutical, Ormond Beach, Florida
  - Clinical Research of Central Florida, Plant City, Florida
  - Accord Clinical Research,LLC, Port Orange, Florida
  - Meridian Research, St. Petersburg, Florida
  - Meridian Research, Tampa, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Mount Vernon Clinical Research, Atlanta, Georgia
  - Gastroenterology Consultants PC, Atlanta, Georgia
  - Atlanta Gastroenterology Assoc, Marietta, Georgia
  - Advanced Digestive Care Center , PC, Stockbridge, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Heartland Research Associates, Newton, Kansas
  - Heartland Research Associates, Wichita, Kansas
  - Research Integrity, Owensboro, Kentucky
  - East Jefferson Gastro, Metairie, Louisiana
  - Boston Clinical Trials Inc, Boston, Massachusetts
  - Beacon Clinical Research, Brockton, Massachusetts
  - Bay State Clinical Trials, Inc., Watertown, Massachusetts
  - Clinical Research Institute, Chesterfield, Michigan
  - Bayer Research, Kalamazoo, Michigan
  - GI Associates and Endoscopy Center, Jackson, Mississippi
  - Quality Clinical Research, Inc, Omaha, Nebraska
  - Central Jersey Medical Research Center, Elizabeth, New Jersey
  - University Hospital,150 Bergen Street,B-134 Pharmacy, Newark, New Jersey
  - Hosc Inc., Brooklyn, New York
  - NY Scientific,189-11 Jamaica Ave, Hollis, New York
  - Peters Medical Research, High Point, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Valley Medical Research, Centerville, Ohio
  - Rapid Medical Research , Inc, Cleveland, Ohio
  - Radiant Research, Columbus, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - Detweiler Family Medicine and Associates, PC, Lansdale, Pennsylvania
  - Clinical Trials Research Services, LLC, Pittsburgh, Pennsylvania
  - Radiant Research, Greer, South Carolina
  - Clinsearch LLC, Chattanooga, Tennessee
  - HCCA-CRS, Jackson, Tennessee
  - KRK Medical Research, Dallas, Texas
  - Gastroenterology Consultants P.A, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Digestive Health Center, Pasadena, Texas
  - Paragon Research Center, San Antonio, Texas
  - Quality Research, Inc, San Antonio, Texas
  - Sun Research, San Antonio, Texas
  - Texas Medical Research Associates , LLC, San Antonio, Texas
  - Breco Research, Sugarland, Texas
  - Pioneer Research Solutions , Inc, Sugarland, Texas
  - Charlottesville Medical Research Center, Charlottesville, Virginia
  - BlueRidge Medical Research, Lynchburg, Virginia
  - Health Research of Hampton Roads, Newport News, Virginia